CLINICAL TRIAL: NCT04996147
Title: Acute and Long-term Impact of Cancer Treatment on Quality-of-life, Physical and Cognitive Function of Head and Neck Cancer Patients
Brief Title: Acute and Long-term Impact of Cancer Treatment on Head and Neck Cancer Patients: FIT4TREATMENT
Acronym: F4T
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government); University Institute of Maia (Other)
Responsible Party: Sponsor
Other Study IDs: 102/2019
Record Dates: First submitted 2021-04-25; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; Acute adverse events; Long-term adverse events; Quality of life; Cognitive function; Physical function
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and Neck Squamous Cell Carcinoma (HNSCC) is the 6th most common cancer. Most cases are diagnosed in locally advanced stages, with treatment involving multimodal approach with combinations of radiotherapy, surgery and chemotherapy. The aggressive nature of HNSCCs and treatment modalities are associated with important acute and late toxicities that often promote temporary or definitive treatment interruption and may compromised the capability to tolerate subsequent treatments. Thus, the aim of this study is to analyze the acute and long-term impact of cancer treatment on quality of life, physical and cognitive function of HNSCC patients diagnosed with a locally advanced disease.

DETAILED DESCRIPTION:
Potential cases will be identified at the multidisciplinary head and neck group meeting. If the case meets eligibility an informed consent will be presented to the patient. Interested participants will be scheduled for baseline assessment before the beginning of treatment (M0). At the end of CRT patients will be submitted to a second assessment (M1). Follow-up assessments will occur 16th to 18th weeks after the treatment is completed (M2). Patients proposed to surgery or induction chemotherapy will also be submitted to an additional assessment before the beginning of CRT (Mc / Mic).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Diagnosis of locally advanced head and neck cancer (oral cavity, oropharynx, hypopharynx, larynx), stage III-IVB.
* Proposed for primary treatment with curative intent - surgery or induction chemotherapy before chemoradiotherapy (CRT) or CRT alone.

Exclusion Criteria:

* Synchronous tumors or other comorbidities with associated uncontrolled symptoms.
* Inability to provide informed consent.
* Expected inability to fulfil the propose schedule and follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients had to have more than 18 years, diagnosed with stage III to IVB HNSCC and proposed for primary treatment with curative intent - surgery or induction chemotherapy before chemoradiotherapy (CRT) or CRT alone. Exclusion criteria was: 1) synchronous tumors or other comorbidities with associated uncontrolled symptoms; 2) inability to provide informed consent; 3) expected inability to fulfil the propose schedule and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Quality of life (acute) | Change of global quality of life score from baseline to the end of treatment
  Global quality of life score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents a high level of functioning)
Quality of life (long-term) | Change of global quality of life score from baseline to 4 months after the treatment is completed
  Global quality of life score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents a high level of functioning)

SECONDARY OUTCOMES:
Fatigue (acute) | Change of fatigue score from baseline to the end of treatment
  Fatigue score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents high level of symptomatology / problems)
Fatigue (long-term) | Change of fatigue score from baseline to 4 months after the treatment is completed
  Fatigue score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents high level of symptomatology / problems)
Social functioning (acute) | Change of body mass index from baseline to the end of treatment
  Social functioning score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents a high level of functioning)
Social functioning (long-term) | Change of body mass index from baseline to 4 months after the treatment is completed
  Social functioning score evaluated by EORTC QLQ-C30 questionnaire (range in score from 0 to 100, high score represents a high level of functioning)
Body composition (acute) | Change of body mass index from baseline to the end of treatment
  Body mass index, evaluated by bioelectrical impedance (BMI kg/m^2).
Body composition (long-term) | Change of body mass index from baseline to 4 months after the treatment is completed
  Body mass index, evaluated by bioelectrical impedance (BMI kg/m^2).
Cognitive function (acute) | Change of MoCA score from baseline to the end of treatment
  Evaluated by the Montreal Cognitive Assessment and the Functional Assessment of Cancer Therapy-Cognitive (MoCA score range between 0 and 30, a score of 26 or over is considered to be normal).
Cognitive function (long-term) | Change of MoCA score from baseline to 4 months after the treatment is completed
  Evaluated by the Montreal Cognitive Assessment and the Functional Assessment of Cancer Therapy-Cognitive (MoCA score range between 0 and 30, a score of 26 or over is considered to be normal).
Dysphagia (acute) | Change of EAT-10 score from baseline to the end of treatment
  Severity of dysphagia assessed by Eating Assessment Tool (EAT-10 total score ranges from 0 to 40, with a score ≥ 3 indicative of dysphagia)
Dysphagia (long-term) | Change of EAT-10 score from baseline to 4 months after the treatment is completed
  Severity of dysphagia assessed by Eating Assessment Tool (EAT-10 total score ranges from 0 to 40, with a score ≥ 3 indicative of dysphagia)
Dysphagia (acute) | Change of FOIS score from baseline to the end of treatment
  Severity of dysphagia assessed by Functional Oral Intake Scale (FOIS ranges from 1 to 7)
Dysphagia (long-term) | Change of FOIS score from baseline to 4 months after the treatment is completed
  Severity of dysphagia assessed by Functional Oral Intake Scale (FOIS ranges from 1 to 7)
Nutritional status (acute) | Change of PG-SGA total score from baseline to the end of treatment
  Evaluated by the Patient-Generated Subjective Global Assessment (PG-SGA range from 0-35 with a higher score reflecting a greater risk of malnutrition).
Nutritional status (long-term) | Change of PG-SGA total score from baseline to 4 months after the treatment is completed
  Evaluated by the Patient-Generated Subjective Global Assessment (PG-SGA range from 0-35 with a higher score reflecting a greater risk of malnutrition).
Handgrip maximal isometric muscle strength (acute) | Change of muscle strength from baseline to the end of treatment
  Measured with manual dynamometers (Kgf).
Handgrip maximal isometric muscle strength (long-term) | Change of muscle strength from baseline to 4 months after the treatment is completed
  Measured with manual dynamometers (Kgf).
Quadriceps maximal isometric muscle strength (acute) | Change of muscle strength from baseline to the end of treatment
  Measured with manual dynamometers (Kgf).
Quadriceps maximal isometric muscle strength (long-term) | Change of muscle strength score from baseline to 4 months after the treatment is completed
  Measured with manual dynamometers (Kgf).
Sit-to-stand test (acute) | Change of repetitions from baseline to the end of treatment
  Sit-to-stand test during 30 seconds
Sit-to-stand test (long-term) | Change of repetitions from baseline to 4 months after the treatment is completed
  Sit-to-stand test during 30 seconds
Physical function (acute) | Change of distance from baseline to the end of treatment
  6 minutes walking test (meters).
Physical function (long-term) | Change of distance from baseline to 4 months after the treatment is completed
  6 minutes walking test (meters)
Progression free survival | 2 years follow-up
  Defined as the time from the beginning of treatment to the date of first progression or death (whichever occurs first) and will be censored at last follow-up date if the patient does not have the event. A progression (local, regional or distant) will be assumed accordingly to the imaging evaluation and/or histopathologic confirmation.
Overall survival | 2 years follow-up
  Defined as the time from the beginning of treatment to the date of death from any cause, for patients who do not die, it will be censored at their last follow-up date.
Capability of tolerating subsequent treatments | 2 years follow-up
  Defined as the proportion of patients that complete the first cycle of the first line palliative chemotherapy after a documented progression (considering all patients with a formal indication).

CONTACTS AND LOCATIONS:
Overall Officials: Inês Leão, MD, Principal Investigator — Centro Hospitalar Vila Nova de Gaia / Espinho
Locations (1):
- Centro Hospitalar Vila Nova de Gaia / Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No